CLINICAL TRIAL: NCT01207219
Title: The Impacts of Yoga and Aerobic Exercise on Neuro-cognitive Function and Symptoms in Early Psychosis - A Single-blind Randomized Controlled Clinical Trial
Brief Title: Yoga and Aerobic Exercise in Psychosis
Acronym: YEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eric Y H Chen, Professor, Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YEP_2010
Record Dates: First submitted 2010-09-16; First posted 2010-09-22 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Psychotic Disorder
Keywords: psychosis; yoga; aerobic exercise; memory; attention; neuro cognition
MeSH Terms: conditions — Psychotic Disorders | interventions — Yoga; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yoga therapy (Experimental): Hatha yoga including breathing control (10 minutes), body posture(40-45minutes), and relaxation (5 minutes).
  Interventions: Behavioral: Yoga therapy
- Aerobic exercise (Experimental): Aerobic exercise includes walking on the treadmill for 15-20 minutes and stationary cycling for 25-30 minutes.
  Interventions: Behavioral: Aerobic exercise
- Waitlist group (No Intervention): Patients in waiting list will be treated as usual and acted as control group.

INTERVENTIONS:
Behavioral: Yoga therapy — 3 sessions per week for 12 weeks, total 36 sessions. Each session lasts around one hour.
  Arms: Yoga therapy
Behavioral: Aerobic exercise — 3 session per week for 12 weeks, total 36 sessions. Each session lasts around one hour.
  Arms: Aerobic exercise

SUMMARY:
The current study aims to evaluate the impacts of yoga and aerobic exercise on neuro-cognitive function, symptoms and brain changes in early psychosis. A total of 120 female subjects who aging from 18-55 years old, and diagnosed with psychotic disorders within the past 5 years, will be randomized into 3 groups: 1) yoga therapy, 2) aerobic exercise, and 3) waitlist group as the control. All groups will try to be kept consistent with their medication with no more than 25% change in their entry level dosage for at least six weeks. The primary outcomes of the present study will be neuro-cognitive changes; the secondary outcomes will be changes of brain structure and function.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND PURPOSE

The present study aims to:

1. Compare the effects of a 12-week integrated yoga therapy and 12-week aerobic exercise program (walking and cycling) on cognitive functions, brain structures and function in female psychosis patients.
2. Compare the changes in physical fitness, clinical symptoms, body-perception, drug adherence, quality of life, and medicational side-effects.

Descriptive data acquired from this study will contribute to a better understanding of the research implications and clinical applications of yoga and aerobic exercise.

SUBJECTS This is a single-blinded, randomized, prospective study using psychopathological assessments, self-rating scales and imaging techniques. In this study, only female psychosis patients will be recruited from the Early Assessment Service for Young People with Psychosis Program (EASY) in Hong Kong, aiming to examine if there is any gender difference in comparison to the study by Pajonk et al. (2007), which selected only male subjects.

Ideally, patients taking Benzodiazepine and anti-depressants will be excluded because of the influence of these drugs on the cognitive test results and hippocampal volume. If it is deemed impractical to completely exclude these patients, all subjects will at least be tried to keep consistent with their antipsychotic dosages, by not permitting more than a 25% change in dose in the first 6 weeks after commencement of the intervention.

According to the data presented in the previous study (F. G. Pajonk et al., 2010), and using the statistical significant level 0.05 and the power 0.80, we calculated the sample size for cognitive assessment is 96 (32 each arm) and for brain imaging the sample required will be 48 (16 each arm) (Noordzij et al., 2010). Considering the drop-out rate will be around 30%, we aim to recruit 120 patients (40 each arm) with half of them (20 each arm) undergoing MRI scanning.

PROCEDURES Subjects will be screened by the clinicians in outpatient units in Hong Kong. They will be asked to sign the consent form when they agree to attend the study. Afterwards, they will be randomly divided into their respective intervention group. Each subject will be given a subject number, which will correspond to the group assignment. There will be two sessions of assessments. In the first session, all 120 subjects will be assessed by an investigator for their cognitive function, severity of symptoms, physical fitness, body-perception, drug adherence, quality of life, and medication side-effects. In the second session, the first 20 subjects recruited into each group will undergo a structural MRI and functional MRI (resting) scan at baseline.

Following the 12-week intervention, the subjects will repeat the same assessments and MRI scan as in the pre-intervention. Patients in waitlist will be provided another 3-month yoga or exercise course according to their willing after the waiting period. All the patients will be followed up for 18 months to assess the long-term effects of both interventions in cognition and symptoms.

For the nature of the study, it is difficult to keep patients blind to group allocation, so that the study can hardly be a double-blinded trial but a single-blinded one. Two investigators will do the yoga training and aerobic exercise without knowing the assessment results. Two research assistants will be well-trained and recruited to do the assessment, and remains blind to treatment allocation.

INTERVENTION PROGRAMS Yoga therapy: The yoga therapy consists of breathing control (10 minutes), body postures (40-45 minutes), and relaxation (5 minutes). The yoga therapy will be carried out three times per week for around 60 minutes at each session. The yoga class will be operated with a size of about 5-10 participants according to the general small-group size with one instructor in the commercial yoga studios in Hong Kong. The body postures used in the present study are designed to cover all body parts to give the body an overall strength and stretching.

Aerobic exercise: The aerobic exercise program will include walking on a treadmill (15-20 minutes), and stationary cycling (25-30 minutes), followed by cool-down stretching afterwards (5 minutes). The aerobic exercise program will also take place three times per week for around 45-55 minutes at each session. The heart rate will be continuously monitored during exercise by a portable recorder aiming to maintain the heart rate in the range of 50-60% of the maximum VO2 value, yielding an exercise exertion level which is considered as a moderate intensity. The aerobic training session will be operated with a size of no more than 10 participants.

Discontiuation: yoga and aerobic exercise will be terminated if the subject reports any uncomfortable symptoms or loses interests in continuing. Discontinuation or non-participation will not affect the usual medical treatment and care, which they receive in the clinical settings.

MEASURES The primary outcomes will be the cognitive tests (memory and attention). Severity of symptoms, physical fitness, and imaging data will be the secondary outcomes. For those patients who drop out during the study will be arranged to an additional assessment session at the withdrawal according to the willingness of the participants. Data of these drop-out patients will be used in the final analysis with the intention-to-treat (ITT) method.

All measurements will be taken at baseline, 12 weeks (upon completion of intervention program) and at 18 months for all 120 subjects. MRI will be carried out at baseline and at 12 weeks for the first 60 subjects recruited.

I. Cognitive Functioning

1. Wechsler Adult Intelligence Scale (WAIS): The current study uses Information sub-test and Digit-Symbol-Coding sub-test.
2. Hong Kong List Learning Test (HKLLT): is a validated Chinese list-learning test (Chan et al., 2000). It provides assessments of the processes and organizational strategies involved in verbal learning.
3. Digit Span Test: is a subtest of the Wechsler Adult Intelligence Scale-Revised. (Wechsler, 1981) It includes digit-span forwards (DF) and digit-span backwards (DB) tests.

3. Letter Cancellation Test: subjects are asked to cancel the letter C and E as quickly as possible. Time, number of error and omission items will be recorded (Lezak, Howieson, & Loring, 1995).

4. Stroop Color and Word Test: Assessment of cognitive flexibility, resistance to interference from outside stimuli, and the ability to suppress a prepotent verbal response. (Stroop, 1935) 5. Subjective Cognitive Impairment Scale (SCIS): A 31-item self-reported questionnaire designed to assess the subjective daily life cognitive impairments in patients with schizophrenia.

II. Magnetic Resonance Imaging (MRI) The first 20 subjects recruited into each group will be scanned using a 3T scanner (Philips Achieva 3-Tesla Quasar). A T1-weighted, MPRAGE sequence (TE=3.2ms, TR=7.5ms, flip angle=7°, FOV 240mm×240 mm) of 155 consecutive slices will be acquired at sagittal view with a voxel size of 1mm×1mm×1 mm. A T2*-weighted EPI sequence will be used for functional magnetic resonance (fMRI) resting (TR/TE=2000/32ms, 32 slices) with a voxel size of 3x3x4mm.

III. Physical Fitness:

1. VO2 max (oxygen consumption): is the maximum capacity of an individual's body to transport and utilize oxygen during incremental exercise, which reflects the physical fitness of the individual.
2. Body Mass Index (BMI).
3. Dual-energy X-Ray Absorptiometry (DXA): assesses the body composition and bone density by passing a very low-level x-ray signal through the body.
4. Sit-and-Reach test: is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles.
5. Standing Balance Test: ask the person to stand on one foot for as long as possible. The test will be conducted with the person having their arms on their waist. Repeat the test on the other leg.
6. Star Excursion Balance Test (SEBT) (Olmsted, Carcia, Hertel, & Shultz, 2002): The SEBT is performed with the subject standing at the center of a grid placed on the floor, with 8 lines extending at 45。 increment from the center of the grid. The subject is asked to maintain a single-leg stance while reaching with the contralateral leg (reach leg) as far as possible along the appropriate vector. The distance from the center of the grid to the touch point is measured in centimeters.

IV. Clinical Assessment

1. Positive and Negative Syndrome Scale (PANSS).
2. Calgary Depression Scale (CDS).

V. Quality of Life The Short Form (36) Health Survey (SF-36).

VI. Body-perception and Drug adherence measure

1. Figure Rating Scale (FRS): there are seven male/female contour drawings, numbered "1" to "7", in increasing body size from left to right. Subjects are asked to choose one figure drawing that most accurately represents the size of their own bodies and then one that represents their desired figure.
2. Cognitive Attitude towards Body Size: subjects are asked whether they think they are: 1) underweight; 2) of normal weight; or 3) overweight.
3. Compliance Rating Scale (CRS): is used to assess medication adherence.
4. Drug Attitude Inventory (DAI-30): assesses the subjects' attitude to the current medication they are taking.

VII. Adverse event No current studies reported any physical or mental artifacts of yoga and aerobic exercise. There is some inherent potential risk of injury in any kind of physical activity. All exercises, both yoga and aerobic exercise, will be increased in a progressive manner to minimize this risk.

The adverse event of the antipsychotics will be assessed by UKU, which is a new comprehensive rating scale for psychotropic drugs and a cross-sectional study of side effects in neuroleptic-treated patients.

STATISTICS The Statistical Package for Social Sciences version 17.0 (SPSS 17.0 statistical package) will be used for the data analysis. Primary outcome variables will be cognition (Hong Kong List Learning Test), and structural imaging data (hippocampal and cingulate cortex volume).

A mixed effects model of repeated measure will be used to compare the changes in cognition and clinical symptoms among the three groups. With mixed effects model, all available data of each subject at each time point will be used (R. Gueorguieva & J. H. Krystal, 2004). This strategy was based on the assumption that data were missing at random (Ralitza Gueorguieva & John H Krystal, 2004).With the unstructured covariance structure (Joe et al., 2009), differences between the three intervention groups over time were assessed with a Group x Time interaction term. Primary outcome measures (HKLLT, Digit Span test, Letter Cancellation test) will be first analyzed by including all three groups. For analyses meeting this criterion of statistical significance, follow-up, the priori comparisons of the active intervention groups with the waitlist group were carried out with the same strategy. All tests will be based on two-sided probabilities set at a significance level of 0.05. The Bonferroni correction procedure will be conducted to adjust for the multiple comparisons among groups.The effect size (Cohen's d) will be calculated as well to compare the therapeutic effects of yoga and aerobic exercise among the three groups.

Image processing and analysis will be carried out with the software packages FSL4.1, Freesurfer 5.1 and SPM8. The primary outcomes of structural MRI data will be the changes of grey matter in hippocampus and prefrontal cortex. The primary outcomes of functional MRI data will be the activity changes in prefrontal cortex and cingulate cortex.

ELIGIBILITY:
Inclusion criteria

* Females aged from 18 to 55.
* Based on the Diagnostic and Statistical Manual (DSM-IV) diagnosed to have schizophrenia, schizoaffective disorder, schizophreniform Psychosis, brief psychotic disorders, psychosis not otherwise specified and delusional disorder. Duration of illness is less than 5 years (including 5 years).
* Cantonese-speaking Chinese.
* Ability to understand the nature of the study and to give an informed consent.
* Fewer than 10 hours of yoga and vigorous aerobic exercise (equivalent to jogging at 10 km/hr) in the previous 3 months.

Exclusion criteria

* Severe physical illness (myocardial infarction, hypertension, fracture, spinal problem), seizure disorders, mental retardation or comorbid substance dependence. Heart rate and blood pressure will be measured at the baseline to exclude the patients with abnormal cardiovascular activities.
* Unstable psychotic symptoms.
* Known pregnancy, or other contraindication to MRI.
* A history of brain trauma or organic brain disease.
* Known history of intellectual disability or special school attendance.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie, JX Lin, PhD, Study Chair — Department of Psychiatry, the University of Hong Kong
Locations (1):
- Department of Psychiatry, LKS Faculty of Medicine, the University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Addington J, Addington D, Gasbarre L. Distractibility and symptoms in schizophrenia. J Psychiatry Neurosci. 1997 May;22(3):180-4. PMID 9183116
- [Background] Duraiswamy G, Thirthalli J, Nagendra HR, Gangadhar BN. Yoga therapy as an add-on treatment in the management of patients with schizophrenia--a randomized controlled trial. Acta Psychiatr Scand. 2007 Sep;116(3):226-32. doi: 10.1111/j.1600-0447.2007.01032.x. PMID 17655565
- [Background] Heyn P, Abreu BC, Ottenbacher KJ. The effects of exercise training on elderly persons with cognitive impairment and dementia: a meta-analysis. Arch Phys Med Rehabil. 2004 Oct;85(10):1694-704. doi: 10.1016/j.apmr.2004.03.019. PMID 15468033
- [Background] Kelley WM, Macrae CN, Wyland CL, Caglar S, Inati S, Heatherton TF. Finding the self? An event-related fMRI study. J Cogn Neurosci. 2002 Jul 1;14(5):785-94. doi: 10.1162/08989290260138672. PMID 12167262
- [Background] Kubesch S, Bretschneider V, Freudenmann R, Weidenhammer N, Lehmann M, Spitzer M, Gron G. Aerobic endurance exercise improves executive functions in depressed patients. J Clin Psychiatry. 2003 Sep;64(9):1005-12. doi: 10.4088/jcp.v64n0905. PMID 14628975
- [Background] Lam LC, Tam CW, Lui VW, Chan WC, Chan SS, Chiu HF, Wong A, Tham MK, Ho KS, Chan WM. Modality of physical exercise and cognitive function in Hong Kong older Chinese community. Int J Geriatr Psychiatry. 2009 Jan;24(1):48-53. doi: 10.1002/gps.2072. PMID 18615844
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Pajonk FG, Wobrock T, Gruber O, Scherk H, Berner D, Kaizl I, Kierer A, Muller S, Oest M, Meyer T, Backens M, Schneider-Axmann T, Thornton AE, Honer WG, Falkai P. Hippocampal plasticity in response to exercise in schizophrenia. Arch Gen Psychiatry. 2010 Feb;67(2):133-43. doi: 10.1001/archgenpsychiatry.2009.193. PMID 20124113
- [Background] Sharma VK, Das S, Mondal S, Goswami U, Gandhi A. Effect of Sahaj Yoga on neuro-cognitive functions in patients suffering from major depression. Indian J Physiol Pharmacol. 2006 Oct-Dec;50(4):375-83. PMID 17402267
- [Background] Whitfield-Gabrieli S, Thermenos HW, Milanovic S, Tsuang MT, Faraone SV, McCarley RW, Shenton ME, Green AI, Nieto-Castanon A, LaViolette P, Wojcik J, Gabrieli JD, Seidman LJ. Hyperactivity and hyperconnectivity of the default network in schizophrenia and in first-degree relatives of persons with schizophrenia. Proc Natl Acad Sci U S A. 2009 Jan 27;106(4):1279-84. doi: 10.1073/pnas.0809141106. Epub 2009 Jan 21. PMID 19164577
- [Derived] Woodward ML, Lin J, Gicas KM, Su W, Hui CLM, Honer WG, Chen EYH, Lang DJ. Medial temporal lobe cortical changes in response to exercise interventions in people with early psychosis: A randomized controlled trial. Schizophr Res. 2020 Sep;223:87-95. doi: 10.1016/j.schres.2020.05.043. Epub 2020 May 30. PMID 32487465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period is from Oct 2010 to Jan 2013 in three outpatient clinics in Hong Kong.
Pre-assignment Details: In order to obtain sufficient imaging data for final analysis, a total of 140 patients were recruited and randomized, 16 of them withdrew before starting intervention. Amongst 124 participants, 9 were excluded from final analysis because of changed diagnosis during study period. 95 of 115 participants completed 12-week study.
Groups:
- Yoga Therapy: Hatha yoga, three sessions per week for 12 weeks, each session lasted around one hour.
- Aerobic Exercise: Included walking and cycling, three times per week for 12 weeks, each session lasted around one hour.
- Waitlist Control Group: Patients in waitlist were treated as usual and acted as the control group.
Period: Overall Study
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Started | 45 | 40 | 39
Included in ITT Analysis | 40 | 37 | 38
Completed | 34 | 29 | 32
Not Completed | 11 | 11 | 7
Not completed — changed diagnosis during study period | 5 | 3 | 1
Not completed — Lost to Follow-up | 6 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group | Total
Number analyzed (Participants) | 40 | 37 | 38 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (6.9) | 23.6 (5.6) | 25.3 (8.2) | 24.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 38 | 115
  Male | 0 | 0 | 0 | 0
Years of education [Mean (Standard Deviation); unit: years] | 11.9 (2.1) | 12.8 (3.2) | 12.3 (2.6) | 12.3 (2.7)
Length of illness [Mean (Standard Deviation); unit: years] | 2.4 (1.9) | 2.5 (2.0) | 1.8 (1.9) | 1.8 (1.9)
Smoking [Number; unit: participants]
  Never smoker | 37 | 32 | 37 | 106
  Past smoker | 0 | 1 | 0 | 1
  Current smoker | 3 | 4 | 1 | 8
Substance abuse [Number; unit: participants]
  No substance abuse | 40 | 37 | 38 | 115
  Substance abuse | 0 | 0 | 0 | 0
Diagnosis [Number; unit: participants]
  Schizophrenia | 21 | 19 | 19 | 59
  Schizoaffective disorder | 4 | 6 | 3 | 13
  Schizophreniform disorder | 0 | 1 | 0 | 1
  Brief psychosis | 1 | 1 | 0 | 2
  Psychosis not otherwise specified | 13 | 8 | 15 | 36
  Delusional disorder | 1 | 2 | 1 | 4
Antipsychotic medication dose, Chlorpromazine (CPZ) [Mean (Standard Deviation); unit: mg/day] — "CPZ-EQ is used here to describe the antipsychotics dose. It is a standard unit representing 100 mg of oral dose of chlorpromazine. Mean dose per day is reported here.
  mg/day | 348 (268) | 301 (245) | 260 (211) | 305 (244)
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: units on a scale] — PANSS total score is computed by summing the scores of positive, negative and general symptom subscores. The range of PANSS total score is from 30 to 210, with higher values representing worse outcome.
  units on a scale | 46.9 (15.8) | 46.8 (16.4) | 45.4 (15.2) | 46.4 (15.7)
Calgary Depression Scale (CDS) total score [Mean (Standard Deviation); unit: units on a scale] — CDS total score is computed by summing the scores of nine items of the scale. The range of CDS total score is from 0 to 27, with higher values representing worse outcome.
  units on a scale | 3.6 (3.4) | 3.4 (4.1) | 3.7 (4.7) | 3.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Verbal Acquisition
Description: Total number of corrected encoded words in the first three trials in the random condition of Hong Kong List Learning test.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: correctly encoded words
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Number analyzed (Participants) | 40 | 37 | 38
correctly encoded words
  Baseline | 22.8 (5.8) | 22.0 (7.8) | 22.7 (7.7)
  12 weeks | 29.5 (6.3) | 28.8 (8.2) | 24.8 (8.2)
Statistical Analysis 1: Comparison: Yoga Therapy vs Aerobic Exercise vs Waitlist Control Group; Data analysis was based on the Intention-to-Treatment (ITT) method. Differences between the three intervention groups over time (baseline and 12 weeks) were assessed with a Group x Time interaction term. A priori comparisons of the active intervention groups with the waitlist group were carried out with the same strategy if analyses including all the three groups meet the criterion of statistical significance (P<0.01); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — The p-value for statistical significance in these analyses was 0.01 adjusted for multiple comparisons; mixed-model analysis with a repeated-measures approach including an unstructured variance matrix

2. Primary Outcome: Verbal Retention
Description: The total number of correctly recalled words after short-term (10 minutes) and long-term (30 minutes) delay in the random condition of Hong Kong List Learning test.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: correctly recorded words
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Number analyzed (Participants) | 40 | 37 | 38
correctly recorded words
  Baseline | 14.9 (5.7) | 15.1 (5.1) | 14.5 (7.0)
  12 weeks | 19.4 (5.9) | 21.0 (7.2) | 16.6 (7.3)

3. Primary Outcome: Working Memory
Description: measured by Digit Span backwards test. In this test, the subject was asked to recall a series of numbers in reverse order. The correctly recalled series were scored as 1, and the test contains 14 sequences of numbers. The range of working memory score is from 0 to 14, with higher values representing better outcome.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Number analyzed (Participants) | 40 | 37 | 38
Scores on a scale
  Baseline | 6.8 (2.7) | 6.8 (2.5) | 7.1 (3.3)
  12 weeks | 8.5 (2.9) | 9.4 (2.9) | 7.7 (2.7)

4. Primary Outcome: Attention and Concentration
Description: measured by Letter Cancellation test Q score. The basic version of the task consists of six 52-character rows in which the target character is randomly interspersed approximately 18 times in each row. Subjects were asked to cancel the letter "C" and "E" as quickly as possible. The time to completion, number of error and omission items were recorded. A "quality of search" index (Q), developed by Geldmacher et al., was applied for the analysis. Q is the ratio of correct number to total number of targets multiplied by the ratio of correct number per second. Higher Q scores represent more efficient performance and better attention and concentration. Q scores could range from 0 (worst possible outcome) to 1 (best possible outcome).
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Correct number per second
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Number analyzed (Participants) | 40 | 37 | 38
Correct number per second
  Baseline | 0.76 (0.14) | 0.71 (0.22) | 0.74 (0.15)
  12 weeks | 0.84 (0.18) | 0.77 (0.19) | 0.73 (0.17)

5. Secondary Outcome: Severity of Symptoms
Description: PANSS total score is computed by summing the scores of positive, negative and general symptom subscores. The range of PANSS total score is from 30 to 210, range of PANSS positive and negative subscores is from 7 to 49, range of PANSS general symptoms subscore is from 16 to 112, with higher values representing worse outcome. CDS total score is computed by summing the scores of nine items of the scale. The range of CDS total score is from 0 to 27, with higher values representing worse outcome.
Time Frame: Baseline and 12 weeks
Population: One subject in the waitlist control group has not completed all measures both at the baseline and 12 weeks. Measure of clinical severity has been missing in the data set. So that there are 37 subjects' data of clinical severity has been included for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Number analyzed (Participants) | 40 | 37 | 37
units on a scale
  PANSS total score-Baseline | 46.9 (15.8) | 46.8 (16.4) | 45.4 (15.2)
  PANSS total score-12 weeks | 37.4 (9.6) | 39.5 (11.1) | 49.0 (15.8)
  PANSS positive subscore-Baseline | 9.9 (3.5) | 9.7 (4.6) | 9.8 (3.8)
  PANSS positive subscore-12 weeks | 8.4 (2.5) | 8.3 (2.5) | 10.0 (3.5)
  PANSS negative subscore-Baseline | 11.0 (4.3) | 11.2 (5.7) | 11.2 (4.1)
  PANSS negative subscore-12 weeks | 8.7 (2.8) | 9.7 (3.8) | 12.6 (5.1)
  PANSS general symptoms-Baseline | 26.0 (9.5) | 25.9 (9.5) | 24.5 (9.2)
  PANSS general symptoms-12 weeks | 20.3 (5.6) | 21.6 (6.9) | 26.4 (9.6)
  CDS-Baseline | 3.6 (3.4) | 3.4 (4.1) | 3.7 (4.7)
  CDS-12 weeks | 1.7 (2.5) | 1.7 (2.4) | 4.3 (4.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: a self-reported questionnaire
Arm/Group | Yoga Therapy | Aerobic Exercise | Waitlist Control Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/45 | 0/40 | 0/39

LIMITATIONS AND CAVEATS:
Lack of a healthy control group; a measurement bias may exist in the HKLLT because the same word list was used for baseline and 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No